CLINICAL TRIAL: NCT04604327
Title: Ensayo clínico Aleatorizado, Abierto, Para Evaluar el Efecto de Dosis profilácticas o terapéuticas de Bemiparina en Pacientes Con COVID-19
Brief Title: Comparison of Two Different Doses of Bemiparin in COVID-19
Acronym: BEMICOP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BEMICOP
Record Dates: First submitted 2020-10-23; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic bemiparin (3,500 IU/day) (Active Comparator): Bemiparin 3,500 IU daily for 10 days
  Interventions: Drug: Bemiparin sodium
- Full therapeutic bemiparin (weight adjusted) (Experimental): Bemiparin at full therapeutic dose, adjusted to body weight, for 10 days
  Interventions: Drug: Bemiparin sodium

INTERVENTIONS:
Drug: Bemiparin sodium — Prophilactic vs full-dose for 10 days
  Other Names: Hibor

SUMMARY:
Patients requiring hospitalization due to COVID-19 pneumonia (non-severe) will be randomized to standard prophylactic doses or full therapeutic dose of bemiparin (a LMWH) for 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Age (equal or more than 18 yo)
* Hospitalization at conventional wards due to COVID-19 related mild or moderate pneumonia (CURB65<3 points; Sat. O2>90%)
* 3-4 points according to the WHO ordinal scale.
* Confirmed COVID-19 (PCR or other validated test)
* D-dimer >500 ng/mL
* Sign of informed consent
* The patient is able, according to investigator's opinion, to deal with all the requirements of the clinical trial.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2020-10-26 (Estimated); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Clinical deterioration | 10 days
  Combined outcome that includes number of patients who suffer any of the following: Death, ICU admission, mechanical ventilatory support, progression to moderate or severe ARDS (according to Berlin criteria) or arterial or venous thrombosis.

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Lecumberri, Md, PhD, Principal Investigator — University of Navarra
Locations (12):
- Spain (12):
  - Hospital Rey Juan Carlos, Móstoles, Madrid
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Clinic, Barcelona
  - Hospital Sant Pau, Barcelona
  - Hospital Universitario Bellvitge, L'Hospitalet de Llobregat
  - Fundación Jiménez Díaz, Madrid
  - Hospital Clínico San carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Complejo Hospitalario de Toledo, Toledo
  - Hospital Universitario Río Hortega, Valladolid

REFERENCES:
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208
- [Derived] Marcos-Jubilar M, Carmona-Torre F, Vidal R, Ruiz-Artacho P, Filella D, Carbonell C, Jimenez-Yuste V, Schwartz J, Llamas P, Alegre F, Sadaba B, Nunez-Cordoba J, Yuste JR, Fernandez-Garcia J, Lecumberri R; BEMICOP Investigators. Therapeutic versus Prophylactic Bemiparin in Hospitalized Patients with Nonsevere COVID-19 Pneumonia (BEMICOP Study): An Open-Label, Multicenter, Randomized, Controlled Trial. Thromb Haemost. 2022 Feb;122(2):295-299. doi: 10.1055/a-1667-7534. Epub 2021 Dec 29. PMID 34638151